CLINICAL TRIAL: NCT04585555
Title: Physiologic Signals and Signatures With the Accuryn Monitoring System - A Retrospective and Prospective Analysis (The Accuryn Registry)
Brief Title: Physiologic Signals and Signatures With the Accuryn Monitoring System (The Accuryn Registry)
Status: Completed | Type: Observational
Sponsor: Potrero Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD-06-2963
Record Dates: First submitted 2020-08-21; First posted 2020-10-14 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Acute Kidney Injury; Abdominal Compartment Syndrome; Intraabdominal Hypertension; Cardiovascular Surgery
MeSH Terms: conditions — Acute Kidney Injury; Intra-Abdominal Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Accuryn Monitoring System: Observational only (no intervention). Patients undergoing cardiovascular surgical intervention(s) monitored with the Accuryn Monitoring System (per standard of care) during their hospital stay.
  Interventions: Device: Accuryn Monitoring System

INTERVENTIONS:
Device: Accuryn Monitoring System — The Accuryn Monitoring System is a novel Foley catheter and monitoring device capable of detecting physiologic changes in vital signs via sensors within the catheter system. These data are captured non-invasively, continuously, and at a high frequency.

SUMMARY:
The Accuryn Registry Study is an open-ended, global, multi-center, retrospective and prospective, single-arm data collection study with an FDA cleared device. The target population are cardiovascular surgery patients. Physiologic data measurements will be collected from enrolled subjects using electronic medical records and data streams via the Accuryn Monitoring System.

DETAILED DESCRIPTION:
The primary objective of the Accuryn Registry Study is to is to track and analyze changes in physiologic data streams using the Accuryn Monitoring System and correlate these changes to the occurrence of acute kidney injury (AKI) following cardiovascular surgery intervention(s).

The secondary objective is to determine the incidence of IAH and ACS in the cardiovascular surgery population and the correlation of these diagnoses to the diagnosis of AKI.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age ≥ 18).
2. Monitored on the Accuryn® Monitoring System during hospital stay.
3. Patient is undergoing cardiovascular surgical intervention(s).

Exclusion Criteria:

1. The patient is unsuitable for the study, in the opinion of the investigator. This may include vulnerable patient populations such as prisoners or those detained in a penal institution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiovascular surgical intervention(s) monitored with the Accuryn Monitoring System (per standard of care) during their hospital stay.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-10-06 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Urine Output (UO) | 30 days
  High accuracy Urine Output (mL/hour) while on a urinary catheter, and estimated UO while not on a urinary catheter
Intra-Abdominal Pressure (IAP) | 30 days
  Intra-Abdominal Pressure (mmHg) trending while on a urinary catheter, as well as active measurements taken by clinician
Temperature (T) | 30 days
  Temperature (degrees Celsius) trending during hospital stay
Intraabdominal Hypertension (IAH) | 30 days
  Intra-abdominal pressure (IAP) above 12 mm Hg (timepoint and duration)
Abdominal Compartment Syndrome (ACS) | 30 days
  Intra-abdominal pressure (IAP) above 20 mm Hg with new organ dysfunction or failure (timepoint and duration)
Acute Kidney Injury (AKI) | 30 days
  % of patients diagnosed with AKI, and hospitalization day of diagnosis. AKI diagnosed per KDIGO criteria (Stage 1 to 3)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Prabhakar, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided